CLINICAL TRIAL: NCT01338467
Title: Glaucoma Treatment by Circular Cyclocoagulation Using High Intensity Focused Ultrasound (HIFU). A Prospective, Multicenter, Open-label, Safety and Efficacy Study of the Treatment With the EYEOP Medical Device in Patients With Refractory Glaucoma
Brief Title: Glaucoma Treatment by Circular Cyclocoagulation Using High Intensity Focused Ultrasound With the EYEOP Medical Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeTechCare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EYEMUST; 2011-A00196-35 (Other: French Health Product Safety Agency (AFSSAPS))
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2013-03

CONDITIONS: Glaucoma
Keywords: Glaucoma; Refractory glaucoma; Cyclocoagulation; High Intensity Focused Ultrasound
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EYEOP Treatment (Experimental): Open label, all subject treated by the EYEOP device
  Interventions: Device: EYEOP device

INTERVENTIONS:
Device: EYEOP device — Cyclocoagulation using High Intensity Focused Ultrasound with EYEOP device

SUMMARY:
The aim of the study is to evaluate the effectiveness and the safety of the EYEOP treatment using High Intensity Focused Ultrasound in refractory glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma included pseudo-exfoliative glaucoma and pigmentary glaucoma in the study eye with maximally tolerated medical treatment
* Ocular hypertension defined as an intraocular pressure (IOP) > 21 mm Hg
* Subject has failed a conventional intraocular glaucoma filtering surgery
* Patient must be aged 18 years or more
* No previous intraocular glaucoma surgery or laser treatment in the study eye during the 3 months before HIFU treatment
* No previous cyclophotocoagulation procedure in the study eye
* Patient able and willing to provide informed consent and to complete post-operative follow-up requirements.

Exclusion Criteria:

* History of previous glaucoma surgery with implantation of glaucoma drainage device in the study eye
* History of ocular or retrobulbar tumor
* Retinal detachment, choroidal hemorrhage or detachment
* Ocular infectious disease within 14 days before HIFU treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Primary efficacy measure : | 6 months
  IOP change (mmHg and Percent) from baseline to 6 months post-HIFU treatment

SECONDARY OUTCOMES:
Safety measures | 6 months
  The incidence of device and procedure-related complications during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DENIS, MD, Principal Investigator — Croix Rousse Hospital - Lyon - France; Laurent FARCY, Study Director — EyeTechCare; Florent APTEL, MD, Principal Investigator — University Hospital - Grenoble - France
Locations (9):
- France (9):
  - University Hospital, Dijon
  - University Hospital, Grenoble
  - University Hospital - Cl Huriez, Lille
  - Clinique du Parc - Private Hospital, Lyon
  - Croix Rousse Hospital, Lyon
  - XV-XX National Ophthalmologic Hospital, Paris
  - XV-XX Ophthalmologic Hospital, Paris
  - Saint-Joseph Hospital, Paris
  - Val de Grace Hospital, Paris

REFERENCES:
- [Result] Denis P, Aptel F, Rouland JF, Nordmann JP, Lachkar Y, Renard JP, Sellem E, Baudouin C, Bron A. Cyclocoagulation of the ciliary bodies by high-intensity focused ultrasound: a 12-month multicenter study. Invest Ophthalmol Vis Sci. 2015 Jan 20;56(2):1089-96. doi: 10.1167/iovs.14-14973. PMID 25604688